CLINICAL TRIAL: NCT03332797
Title: A Phase Ia/Ib, Multicenter, Open-Label, Dose Escalation, Dose Expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-9545 Alone or in Combination With Palbociclib and/or LHRH Agonist in Patients With Locally Advanced or Metastatic Estrogen Receptor-Positive Breast Cancer
Brief Title: A Study of GDC-9545 Alone or in Combination With Palbociclib and/or Luteinizing Hormone-Releasing Hormone (LHRH) Agonist in Locally Advanced or Metastatic Estrogen Receptor-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO39932; 2017-002083-41 (EudraCT Number); 2023-506700-12-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; palbociclib; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Dose Escalation: GDC-9545 (Experimental): During dose escalation, postmenopausal participants will be assigned sequentially to escalating doses of GDC-9545, up to the maximum tolerated dose (MTD) or maximum administered dose (MAD).
  Interventions: Drug: GDC-9545
- Dose Escalation: Cohort B0: GDC-9545 + Palbociclib (Experimental): GDC-9545 will be administered to postmenopausal participants, at a dose lower than the MTD or MAD determined in single-agent dose escalation, in combination with the label-recommended dose of palbociclib.
  Interventions: Drug: GDC-9545; Drug: Palbociclib
- Dose Expansion: Cohort A1: GDC-9545 Dose 1 (Experimental): GDC-9545 will be administered to postmenopausal participants as a single-agent at a dose that is less than or equal to the MTD/MAD (Dose 1).
  Interventions: Drug: GDC-9545
- Dose Expansion: Cohort A2: GDC-9545 Dose 1 + LHRH (Experimental): GDC-9545 will be administered to pre- or perimenopausal participants at a dose that is less than or equal to the MTD/MAD (Dose 1) in combination with an approved LHRH agonist.
  Interventions: Drug: GDC-9545; Drug: LHRH Agonist
- Dose Expansion: Cohort A3: GDC-9545 Dose 2 (Experimental): GDC-9545 will be administered to postmenopausal participants as a single-agent at a dose that is less than or equal to the MTD/MAD (Dose 2).
  Interventions: Drug: GDC-9545
- Dose Expansion: Cohort A4: GDC-9545 Dose 2 + LHRH (Experimental): GDC-9545 will be administered to pre- or perimenopausal participants at a dose that is less than or equal to the MTD/MAD (Dose 2) in combination with an LHRH agonist.
  Interventions: Drug: GDC-9545; Drug: LHRH Agonist
- Dose Expansion: Cohort A5: GDC-9545 Dose 3 (Experimental): GDC-9545 will be administered to postmenopausal participants as a single-agent at a dose that is less than or equal to the MTD/MAD (Dose 3).
  Interventions: Drug: GDC-9545
- Dose Expansion: Cohort B1: GDC-9545 + Palbociclib (Experimental): GDC-9545 will be administered to postmenopausal participants, at a dose that is less than or equal to the MTD/MAD, in combination with the label-recommended dose of palbociclib.
  Interventions: Drug: GDC-9545; Drug: Palbociclib
- Dose Expansion: Cohort B2: GDC-9545 + Palbociclib + LHRH (Experimental): GDC-9545 will be administered to pre- or perimenopausal participants, at a dose that is less than or equal to the MTD/MAD, in combination with the label-recommended dose of palbociclib and an approved LHRH agonist.
  Interventions: Drug: GDC-9545; Drug: Palbociclib; Drug: LHRH Agonist
- Dose Expansion: Cohort C1: GDC-9545 Dose 2 +/- Palbociclib (Experimental): GDC-9545 will be administered to postmenopausal participants at a pre-defined dose level (Dose 2) as a single agent for 14 days, followed by treatment with either GDC-9545 (Dose 2) plus palbociclib or GDC-9545 (Dose 2) alone for the duration of the study, as determined by the investigator.
  Interventions: Drug: GDC-9545; Drug: Palbociclib
- Dose Expansion: Cohort C2: GDC-9545 Dose 2 + Palbociclib (Experimental): GDC-9545 will be administered to postmenopausal participants at a pre-defined dose level (Dose 2), in combination with the label-recommended dose of palbociclib.
  Interventions: Drug: GDC-9545; Drug: Palbociclib
- Dose Expansion: Cohort X: GDC-9545 Dose 3 (Experimental): GDC-9545 will be administered at a pre-defined dose level (Dose 3) to postmenopausal participants currently receiving clinical benefit with GDC-0927 or GDC-0810 on Studies GO29656 (NCT02316509) or GO29642 (NCT01823835), respectively, upon completion of their studies.
  Interventions: Drug: GDC-9545

INTERVENTIONS:
Drug: GDC-9545 — GDC-9545 will be administered orally, once daily, on Days 1-28 of each 28-day cycle, until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Giredestrant; RO7197597; RG6171
Drug: Palbociclib — Palbociclib will be administered orally, once daily, at the label-recommended dose of 125 mg on Days 1-21 of each 28-day cycle, until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Arms: Dose Escalation: Cohort B0: GDC-9545 + Palbociclib; Dose Expansion: Cohort B1: GDC-9545 + Palbociclib; Dose Expansion: Cohort B2: GDC-9545 + Palbociclib + LHRH; Dose Expansion: Cohort C1: GDC-9545 Dose 2 +/- Palbociclib; Dose Expansion: Cohort C2: GDC-9545 Dose 2 + Palbociclib
Drug: LHRH Agonist — The LHRH agonist (leuprolide acetate, goserelin acetate, or triptorelin pamoate) will be administered by injection once every 4 weeks on Day 1 of each 28-day cycle, according to the label. The investigator will choose the appropriate LHRH agonist approved for use in breast cancer.
  Arms: Dose Expansion: Cohort A2: GDC-9545 Dose 1 + LHRH; Dose Expansion: Cohort A4: GDC-9545 Dose 2 + LHRH; Dose Expansion: Cohort B2: GDC-9545 + Palbociclib + LHRH

SUMMARY:
This study will evaluate the safety, pharmacokinetic (PK), pharmacodynamic (PD) activity, and preliminary anti-tumor activity of GDC-9545 as a single agent and in combination with palbociclib and/or luteinizing hormone-releasing hormone (LHRH) agonist in participants with advanced or metastatic estrogen receptor (ER)-positive (human epidermal growth factor receptor 2 [HER2]-negative) breast cancer.

ELIGIBILITY:
Inclusion Criteria for Dose Escalation:

* Histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of either locally recurrent disease not amenable to resection or radiation therapy with curative intent or with metastatic disease
* Estrogen receptor (ER)-positive tumor
* Human epidermal growth factor receptor 2 (HER2)-negative breast cancer as per local laboratory testing
* Measurable disease, or evaluable bone disease; that is, bone lesions that are lytic or mixed (lytic + sclerotic) in the absence of measurable lesion
* Required paired pre- and on-treatment tumor biopsies for participants with metastases that are safely accessible as determined by the investigator
* Advanced or metastatic ER-positive/HER2-negative breast cancer that has recurred or progressed while being treated with adjuvant endocrine therapy for a duration of at least 24 months and/or endocrine therapy in the incurable, locally advanced, or metastatic setting and derived a clinical benefit from therapy (i.e., tumor response or stable disease for at least 6 months)
* No more than 2 prior lines of treatment for advanced or metastatic breast cancer
* Greater than or equal to (≥)2 weeks must have elapsed from the use of any other endocrine, targeted therapy or chemotherapy
* Single-Agent Cohorts (only applies to Dose Escalation): Advanced or metastatic disease that is either refractory to or intolerant of existing standard therapy or for which no effective standard therapy that confers clinical benefit is available
* Cohort B0: No prior treatment with cyclin-dependent kinase 4/6 (CDK4/6) inhibitor
* For participants undergoing 18F-fluoroestradiol-positron emission tomography (FES-PET) imaging additional restrictions on prior therapy include: ≥2 months must have elapsed from the use of tamoxifen; ≥6 months must have elapsed from the use of fulvestrant
* Postmenopausal status
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (≤)1
* Resolution of all acute toxic effects of prior therapy or surgical procedures to baseline or Grade ≤1 (except alopecia or other toxicities not considered to be a safety risk for the patient)
* Life expectancy of ≥12 weeks
* Adequate organ function

Inclusion Criteria for Dose Expansion:

Same criteria as above for Dose Escalation, except for those that only apply to Dose Escalation, plus the following:

* Required paired pre- and on-treatment tumor biopsies for participants in Cohorts A1-A5, B1, and B2 with metastases that are safely accessible as determined by the investigator
* In South Korea: Must have received exactly 2 prior lines of treatment for advanced or metastatic breast cancer
* In the rest of the world: No more than 1 prior line of treatment for advanced or metastatic breast cancer (not applicable to Cohort X)

Plus the following criteria:

* Cohorts B1 and B2: No prior treatment with CDK4/6 inhibitor
* Cohorts A1, A3, A5, B1, C1, and C2 only: Postmenopausal status
* Cohorts A2, A4, and B2 only: Participants not defined as postmenopausal; Age less than (<)56 years who have medical menopause on LHRH agonist (on stable dose ≥4 weeks)
* No prior treatment with an oral selective estrogen receptor degrader (SERD)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods with a failure rate of <1% per year during the treatment period and for 10 days after the last dose of GDC-9545 and 21 days after the last dose of palbociclib, and agreement to refrain from donating eggs during this same period
* Cohort X only: Participants enrolled on Studies GO29656 or GO29642 and received clinical benefit from GDC-0927 or GDC-0810
* Hematology, chemistry, and urinalysis collected 72 hours before Cycle 1, Day 1 deemed acceptable for dosing by the investigator
* No other endocrine therapy, targeted therapy, or chemotherapy after last dose of GDC-0927 or GDC-0810

Exclusion Criteria for Dose Escalation:

* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* Current treatment with any systemic anti-cancer therapies for advanced disease (not applicable to Cohort X participants currently receiving GDC-0810 or GDC-0927)
* Concurrent treatment with warfarin or phenytoin
* Diagnosis of any secondary malignancy within 3 years prior to enrollment, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, or major upper gastrointestinal (GI) surgery including gastric resection
* Known human immunodeficiency virus (HIV) infection
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis (e.g., hepatitis B or hepatitis C virus), current alcohol abuse, or cirrhosis
* Major surgery within 4 weeks prior to enrollment
* Radiation therapy within 2 weeks prior to enrollment
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Inability or unwillingness to swallow tablets or capsules (only applies to Dose Escalation)
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study (only applies to Dose Escalation)
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction
* QT interval corrected using Fridericia's formula (QTcF) greater than (>)470 milliseconds (ms) demonstrated by at least two ECGs >30 minutes apart
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease coronary heart disease clinically significant electrolyte abnormalities or family history of sudden unexplained death or long QT syndrome
* Current treatment with medications that are well known to prolong the QT interval

Exclusion Criteria for Dose Expansion:

Same criteria as above for Dose Escalation, except for those that only apply to Dose Escalation, plus the following criteria:

* Pregnant, lactating, or breastfeeding
* Additional exclusion criteria for Cohort B (Phase 1b cohort): History of venous thromboembolic event requiring therapeutic anticoagulation
* Additional exclusion criteria for Cohorts C1 and C2 only: Current treatment with medications that are well known to decrease heart rate, including beta blockers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE v4.0) | From Baseline until 28 days after the last dose of study treatment (up to 84 months)
Dose Escalation: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of GDC-9545 When Administered as a Single Agent or in Combination with Palbociclib | Days -7 to 28 of Cycle 1
Dose Escalation: Number of Participants with Dose-Limiting Toxicities When GDC-9545 is Administered as a Single Agent or in Combination with Palbociclib | Days -7 to 28 of Cycle 1
Change from Baseline in Systolic Blood Pressure Over Time | Baseline and at each treatment cycle (1 cycle is 28 days) through to 28 days after the last dose of study treatment
Change from Baseline in Diastolic Blood Pressure Over Time | Baseline and at each treatment cycle (1 cycle is 28 days) through to 28 days after the last dose of study treatment
Change from Baseline in Body Temperature Over Time | Baseline and at each treatment cycle (1 cycle is 28 days) through to 28 days after the last dose of study treatment
Change from Baseline in Pulse Rate Over Time | Baseline and at each treatment cycle (1 cycle is 28 days) through to 28 days after the last dose of study treatment
Change from Baseline in Respiration Rate Over Time | Baseline and at each treatment cycle (1 cycle is 28 days) through to 28 days after the last dose of study treatment
Change from Baseline in Electrocardiogram (ECG) Results Over Time: Heart Rate | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Change from Baseline in ECG Results Over Time: PR Duration | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Change from Baseline in ECG Results Over Time: QRS Duration | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Change from Baseline in ECG Results Over Time: QT Duration | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Change from Baseline in ECG Results Over Time: QTcF Duration | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Change from Baseline in ECG Results Over Time: RR Duration | Baseline and at predefined intervals from Cycle 1 and at each subsequent cycle (1 cycle is 28 days) through to the last dose of study treatment
Number of Participants with Clinical Laboratory Abnormalities in Hematology Tests by Highest Grade According to NCI-CTCAE v4.0 | Baseline, Cycle 1, and at each subsequent cycle (1 cycle is 28 days) or at every other cycle starting from Cycle 3 (Cohort X only), up to 28 days after the last dose of study treatment
  Laboratory parameters for hematology will be measured and compared with a standard reference range. Values outside of the standard reference range are considered abnormalities. Not every laboratory abnormality qualifies as an adverse event. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment, a medical intervention, or a change in concomitant therapy; or is clinically significant in the investigator's judgment.
Number of Participants with Clinical Laboratory Abnormalities in Blood Chemistry Tests by Highest Grade According to NCI-CTCAE v4.0 | Baseline, Cycle 1, and at each subsequent cycle (1 cycle is 28 days) or at every other cycle starting from Cycle 3 (Cohort X only), up to 28 days after the last dose of study treatment
  Laboratory parameters for blood chemistry will be measured and compared with a standard reference range. Values outside of the standard reference range are considered abnormalities. Not every laboratory abnormality qualifies as an adverse event. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment, a medical intervention, or a change in concomitant therapy; or is clinically significant in the investigator's judgment.
Number of Participants with Clinical Laboratory Abnormalities in Urinalysis Tests by Highest Grade According to NCI-CTCAE v4.0 | Baseline, Cycle 3, and at every other cycle (1 cycle is 28 days) up to 28 days after the last dose of study treatment
  Laboratory parameters for urinalysis will be measured and compared with a standard reference range. Values outside of the standard reference range are considered abnormalities. Not every laboratory abnormality qualifies as an adverse event. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment, a medical intervention, or a change in concomitant therapy; or is clinically significant in the investigator's judgment.

SECONDARY OUTCOMES:
Plasma Concentration of GDC-9545 Over Time | At predefined intervals from Cycle 1, Day -7 (Single-Agent Dose Escalation and A1-A5 only) or Cycle 1, Day 1 (B0, B1, and B2) to Cycle 4, Day 1 (1 cycle is 28 days) and at study completion; Cycle 1, Days -7 or 8 (C1 only); Cycle 1, Day 8 (C2 only)
Plasma Concentration of Palbociclib Over Time | At predefined intervals from Cycle 1, Day 1 to Cycle 4, Day 1 (1 cycle is 28 days) and at study completion (B0, B1, and B2 only); Cycle 1, Day 8 (C2 only)
Plasma Concentration of LHRH Over Time | At predefined intervals from Cycle 1, Day 1 to Cycle 4, Day 1 (1 cycle is 28 days) and at study completion (B2 only)
Percentage of Participants with Objective Response | For all cohorts, except for Cohort X: Baseline and every 8 weeks from Cycle 1, Day 1 until end of study treatment (up to 84 months)
  Objective response is defined as a complete response or partial response on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1).
Clinical Benefit Rate | For all cohorts, except for Cohort X: Baseline and every 8 weeks from Cycle 1, Day 1 until end of study treatment (up to 84 months)
  Clinical benefit rate is defined as the percentage of participants achieving either of the following: confirmed complete response or partial response (as determined by the investigator according to RECIST v1.1); or the first occurrence of progressive disease after 24 weeks of study treatment.
Duration of Response | For all cohorts, except for Cohort X: From the first occurrence of a documented objective response until first observation of disease progression or death from any cause on study, whichever occurs first (up to 84 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (6):
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- South Korea (5):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Centro Oncologioco MD Anderson Internacional, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - The Royal Marsden Hospital, Suttton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malhi V, Agarwal P, Gates MR, Liu L, Wang J, De Bruyn T, Lam S, Eng-Wong J, Perez-Moreno P, Chen YC, Yu J. Optimizing Early-stage Clinical Pharmacology Evaluation to Accelerate Clinical Development of Giredestrant in Advanced Breast Cancer. Cancer Res Commun. 2023 Dec 15;3(12):2551-2559. doi: 10.1158/2767-9764.CRC-23-0324. PMID 38019116
- [Derived] Jhaveri KL, Bellet M, Turner NC, Loi S, Bardia A, Boni V, Sohn J, Neilan TG, Villanueva-Vazquez R, Kabos P, Garcia-Estevez L, Lopez-Miranda E, Perez-Fidalgo JA, Perez-Garcia JM, Yu J, Fredrickson J, Moore HM, Chang CW, Bond JW, Eng-Wong J, Gates MR, Lim E. Phase Ia/b Study of Giredestrant +/- Palbociclib and +/- Luteinizing Hormone-Releasing Hormone Agonists in Estrogen Receptor-Positive, HER2-Negative, Locally Advanced/Metastatic Breast Cancer. Clin Cancer Res. 2024 Feb 16;30(4):754-766. doi: 10.1158/1078-0432.CCR-23-1796. PMID 37921755